CLINICAL TRIAL: NCT07105280
Title: Closed-Loop Therapeutic Refinement Using Local Field Potentials in Parkinson's Disease
Acronym: CTRL-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HagaZiekenhuis (Other)
Collaborators: Maastricht University Medical Center (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Maria Fiorella Contarino, Principal Investigator, HagaZiekenhuis
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTRL-PD study
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: deep brain stimulation; adaptive therapy; closed-loop therapy; local field potentials; subhtalamic nucleus; parkinson's disease

STUDY DESIGN:
Intervention Model Description: An N-of-1 trial design in which each patient tests conventional DBS, optimized conventional DBS, and optimized adaptive DBS for seven days each, in a blinded and randomized sequence.
Masking Description: Patients are not masked for the group they are in, but they are blinded for the order in which they receive treatment with three different deep brain stimulation settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-of-1 study arm (Experimental): Main study arm where each participant tests conventional DBS, optimized conventional DBS, and optimized adaptive DBS for seven days each, in a blinded and randomized sequence
  Interventions: Device: Conventional DBS; Device: Optimized conventional DBS; Device: Optimized adaptive DBS

INTERVENTIONS:
Device: Conventional DBS — Treatment for a minimum of 2 to a maximum of 7 days with the patient's original conventional DBS (cDBS) settings.
Device: Optimized conventional DBS — Treatment for a minimum of 2 to a maximum of 7 days with a previously optimized version of the patient's original conventional DBS (O-cDBS) settings.
Device: Optimized adaptive DBS — Treatment for a minimum of 2 to a maximum of 7 days with previously optimized adaptive DBS (O-aDBS) settings.

SUMMARY:
This multi-center pilot study compares conventional DBS (cDBS) and adaptive DBS (aDBS) in Parkinson's disease patients using the Medtronic Percept™ system.

The aim of the study is to identify which patients benefit most from aDBS, and to explore patient and LFP signal characteristics as well as stimulation parameters as potential predictors of treatment preference and efficacy. The study utilizes a blinded, randomized N-of-1 trial design, where each patient tests the following:

* Original cDBS settings (cDBS);
* Optimized cDBS settings (O-cDBS);
* Optimized aDBS settings (O-aDBS) Each setting is evaluated for a minimum of 2 and maximum of 7 days at home in a randomized order (patient blinded).

The main study outcome consists of the patient's final preference among the three DBS programs: original cDBS, O-cDBS, or O-aDBS. Secondary outcomes focus on differences between cDBS, O-cDBS and O-aDBS regarding the following parameters (among others):

* Quality of life (PDQ-39);
* Patient satisfaction (5-point Likert Scale);
* (Non)-motor fluctuations (MDS-UPDRS-III + MDS-NMS-Q);
* Time spent in "ON"/"OFF" motor phases (symptom diary + MDS-UPDRS IV);
* Time spent experiencing dyskinesia (symptom diary + MDS-UPDRS IV);
* Time spent with the most bothersome symptom (symptom diary + MDSUPDRS IV);
* Stimulation parameters;
* Local field potentials.

The study also incorporates real-world home-based assessments using the Experience Sampling Method (ESM) to capture motor and non-motor symptom fluctuations in daily life and identify differences among the three settings.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the subthalamic nucleus (STN) is an established treatment for patients with Parkinson's disease (PD), particularly for those experiencing motor fluctuations that do not respond adequately to medication. Optimal clinical outcomes depend on precise programming of stimulation parameters to effectively reduce motor symptoms, while avoiding side effects by minimizing stimulation of adjacent brain structures. During surgery, an electrode with eight contact points (1-3-3-1 design) is permanently implanted.

At the Haga Teaching Hospital, Maastricht UMC+, and Amsterdam UMC, the Medtronic Percept™ PC/RC system is commonly used for PD patients. This system provides not only stimulation but also the ability to record brain signals in the form of local field potentials (LFPs). This recording functionality can offer valuable insights for clinicians to fine-tune DBS parameters. For instance, elevated beta activity (13-35 Hz) in LFPs has been shown to correlate with the severity of symptoms such as rigidity and bradykinesia in PD patients.

In January 2025, a software update was introduced for the Percept™ system, enabling more advanced LFP measurements. This update allows the system to deliver adaptive DBS (aDBS), in which brain signals are used in real-time to continuously and automatically adjust stimulation amplitude. Although aDBS is a promising advancement, comprehensive research comparing its benefits and drawbacks to conventional DBS (cDBS) is still lacking. The only major study, ADAPT-PD, found that aDBS and cDBS result in similar durations of time spent in the "ON" phase, but it did not clarify which subgroup of patients benefits most from aDBS. Interestingly, many participants in the ADAPT-PD study expressed a desire to switch from cDBS to aDBS after the trial, though the factors influencing these preferences remain unclear. This highlights the need for detailed investigation into the relative advantages of aDBS and for whom the current form of aDBS provides the greatest benefit.

This study targets PD patients who have undergone cDBS for at least six months but are not experiencing optimal results due to persistent motor symptoms or stimulation-induced side effects that are insufficiently addressed by standard cDBS. Within this pilot study, using a combined N-of-1 trial design, outcomes of the patient's current cDBS settings and optimized conventional DBS (O-cDBS) will be objectively compared with those of optimized adaptive DBS (O-aDBS).

In an N-of-1 trial, an individual patient undergoes different test and placebo treatments in a randomized order. By conducting multiple N-of-1 trials across several patients, reliable and objective outcomes can be gathered both at the individual and population levels. In this study, each patient will test all three stimulation programs (current cDBS, O-cDBS, and O-aDBS) in a blinded and randomized sequence, each for seven days. The final outcome will be the patient's preferred program, with the patient's personal choice taking priority. To better understand the impact of switching from cDBS to aDBS-and to include effects on patient quality of life-this study will analyze not only motor symptoms but also cognitive and behavioral effects in daily life. This will be assessed through structured questionnaires, including a symptom diary and questions via the Experience Sampling Method (ESM). ESM is a validated, CE-certified digital diary method where patients provide feedback on the patient's symptoms at semi-random times, helping to reduce recall bias. By objectively analyzing the pros and cons of switching from cDBS to aDBS in these specific patient groups, this study aims to support neurologists in the clinical use of this new technology. Furthermore, the findings may contribute to more effective use of the system and ultimately to improved DBS treatment and quality of life for patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease with bilateral DBS in the STN
* DBS surgery with implantation of the Percept™ PC/RC system performed at least 6 months ago
* Symptoms such as dysarthria, freezing, or ON-OFF fluctuations that are insufficiently controlled
* A usable LFP signal is present on at least one side

Exclusion Criteria:

* Patients for whom switching to aDBS, operating the remote control independently, or making regular visits to the DBS center is deemed clinically unsafe or unreliable by the treating physician - for example, due to active or unstable cognitive or psychiatric conditions.
* High impedance, defective DBS electrodes, or insufficient LFP signal quality, or bilateral stimulation primarily on the most ventral or dorsal contact points, preventing proper functioning of aDBS.
* Patients who have objected to the use of their electronic health record data for medical scientific research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient preference of DBS settings | after the three week trial phase of the study
  The patient's choice for one of the three program options (standard cDBS, O-cDBS, or O-aDBS)

SECONDARY OUTCOMES:
Quality of life per DBS settings | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  The 39 item Parkinson's Disease Questionnaire (PDQ-39) score for cDBS, O-cDBS, O-aDBS (score between 0 (good quality) and 100 (bad quality))
General Prompt Experience Sampling Method score per DBS settings | Reported average daily score within each week with one of the DBS settings (at 1-7 days, 8-14 days and 15-21 days)
  Custom general prompt daily (non-)motor fluctuations questionnaire via Experience Sampling Method (ESM), with a score ranging from 0 (good) to 270 (poor)
Patient satisfaction per DBS settings | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  5-point Likert scale score for patient satisfaction with cDBS, O-cDBS and O-aDBS (1=very dissatisfied; 2= dissatisfied; 3=neutral; 4=satisfied; 5=very satisfied)
Time spent in ON/OFF per DBS settings according to symptom diary | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time spent in OFF during time awake for cDBS, O-cDBS and O-aDBS according to symptom diary (0% (good) to 100% (poor)).
Time spent with dyskinesia per DBS setting according to symptom diary | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time awake spent with dyskinesia for cDBS, O-cDBS and O-aDBS according to symptom diary (0% (good), 100% (poor)).
Time spent with most bothersome symptom per DBS setting according to symptom diary | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time awake spent with most bothersome symptom for cDBS, O-cDBS and O-aDBS according to symptom diary. (0% (good), 100% (poor))
Total score for motor fluctuations per DBS setting | Reported at baseline and after optimizing each intervention
  Motor score according to Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS-III) for cDBS, O-cDBS and O-aDBS, with the score ranging from 0 (good) to 132 (poor)
Levodopa equivalent daily dose per DBS setting | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  According to latest levodopa equivalent daily dose scheme, determined for cDBS, O-cDBS and O-aDBS
Time spent in ON/OFF per DBS settings | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time spent in OFF during time awake for cDBS, O-cDBS and O-aDBS according to Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part IV (MDS-UPDRS-IV) for cDBS, O-cDBS and O-aDBS (0% (good) to 100% (poor)).
Time spent with dyskinesia per DBS setting | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time awake spent with dyskinesia for cDBS, O-cDBS and O-aDBS according to Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part IV (MDS-UPDRS-IV) (0% (good), 100% (poor))
Time spent with most bothersome symptom per DBS setting | Reported after each week with one of the DBS settings (at 7 days, 14 days and 21 days)
  Percentage of time awake spent with most bothersome symptom for cDBS, O-cDBS and O-aDBS according to Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part IV (MDS-UPDRS-IV) in case of symptom being either "Motor fluctuations", "Dyskinesia", "OFF- dystonia", (0% (good), 100% (poor)).
Total score for non-motor fluctuations per DBS setting | Reported at baseline and after optimizing each intervention
  Non-motor score according to Movement Disorder Society - Non-Motor Symptom Questionnaire (MDS-NMS-Q) for cDBS, O-cDBS and O-aDBS, with scores ranging from 0 (good) to 208 (poor)).
Morning Prompt Experience Sampling Method score per DBS settings | Reported average daily score within each week with one of the DBS settings (at 1-7 days, 8-14 days and 15-21 days)
  Custom morning prompt daily (non-)motor fluctuations questionnaire via Experience Sampling Method (ESM), with a score ranging from 0 (good) to 35 (poor)
Evening Prompt Experience Sampling Method score per DBS settings | Reported average daily score within each week with one of the DBS settings (at 1-7 days, 8-14 days and 15-21 days)
  Custom evening prompt daily (non-)motor fluctuations questionnaire via Experience Sampling Method (ESM), with a score ranging from 0 (good) to 76 (poor)

OTHER OUTCOMES:
Cognitive functioning at baseline | prior to or at study start (no more than 6 months old)
  Montreal Cognitive Assessment (MoCA) score at baseline (no more than 6 months old), with a score ranging from 0 (poor) to 30 (good).
Disease duration at baseline | at baseline (start of study participation)
  Disease duration in years at baseline (study start)
Age at baseline | at baseline (start of study participation)
  Age in years at baseline (study start)
Biological sex | at baseline (start of study participation)
  Biologically determined sex at baseline
Time after lead implantation at baseline | at baseline (start of study participation)
  Time after lead implantation surgery in months at baseline (study start)
At-home recorded local field potentials per DBS setting | Recorded during each week per DBS setting (1-7 days, 8-14 days, and 15-21 days)
  Local field potentials recorded using BrainSense Timeline and Events for cDBS, O-cDBS and O-aDBS
In-clinic general local field potential recordings | at baseline (start of study participation)
  Local field potential recordings using the BrainSense Survey, Electrode identifier, Setup during in-clinic visit at baseline.
In-clinic local field potential recordings per DBS setting | At baseline and after optimization of each of the DBS settings
  Local field potential recordings using the BrainSense Streaming during in-clinic visits for cDBS, O-cDBS and O-aDBS
Stimulation settings per DBS setting | At the start of each intervention period (at 1 day, 8 days, 15 days)
  Stimulation settings (contact point, power, pulse width, frequency, adaptive protocol (i.e. single or dual threshold + thresholds))

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fiorella Contarino, MD, PhD, Principal Investigator — HagaZiekenhuis
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Maastricht UMC+, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided
Personal data security issues

REFERENCES:
- [Background] Bronte-Stewart H, Beudel M, Ostrem J, Little S, Almeida L, Zamora AR, et al. Chronic Adaptive DBS Provides Similar "On" Time with Trend of Improvement Compared to Continuous DBS in Parkinson's Disease and 98% of Participants Chose to Remain on aDBS (S2.008). Neurology (internet). 2024 Apr 9;102(17_supplement_1). Available from: https://doi.org/10.1212/wnl.0000000000204762
- [Background] Nakajima A, Shimo Y, Fuse A, Tokugawa J, Hishii M, Iwamuro H, Umemura A, Hattori N. Case Report: Chronic Adaptive Deep Brain Stimulation Personalizing Therapy Based on Parkinsonian State. Front Hum Neurosci. 2021 Aug 13;15:702961. doi: 10.3389/fnhum.2021.702961. eCollection 2021. PMID 34483867
- See also: Description Medtronic Percept System (conventioal/adaptive DBS system used in this research) — https://europe.medtronic.com/xd-en/healthcare-professionals/products/neurological/deep-brain-stimulation-systems/percept-pc.html